CLINICAL TRIAL: NCT06105580
Title: Conduction System Pacing vs Biventricular Resynchronization Therapy in Systolic Dysfunction and Wide QRS: Mortality, Heart Failure Hospitalization or Cardiac Transplant
Brief Title: Conduction System Pacing vs Biventricular Pacing in Systolic Dysfunction and Wide QRS: Mortality, Heart Failure Hospitalization or Cardiac Transplant
Acronym: CONSYST-CRT II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Responsible Party: Principal Investigator, Josep Lluis Mont Girbau, Head of Arrhythmia Research., Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CONSYST-CRT II
Record Dates: First submitted 2023-10-04; First posted 2023-10-27 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Resynchronization Therapy; Heart Failure
Keywords: left bundle branch pacing; biventricular pacing; cardiac resynchronization therapy
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Intervention Model Description: The first 130 patients have been recruited in the context of the CONSYST I study (ClinicalTrials.gov Identifier: NCT05187611).
  It is planned to perform an interim analysis (intermediate analysis) for the primary endpoint in all randomized patients who received intervention. The formal limits of stopping the study will be determined by the limits of futility and effectiveness defined by the rules of sequential stopping using the O'Brien-Fleming method. The interim analysis will be performed with a sample recruitment of 50%. Members of the Data Monitoring Committee, but not any trial investigator, will be informed of the results of the interim analysis. A p of 0.0054 (two-sided alpha) will be required for the interim analysis and 0.049 in the final analysis.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conduction system pacing (Experimental): Pacing the His-Purkinje system.
  Crossover to biventricular pacing allowed in case of failed conduction system pacing: failed His bundle pacing and failed Left bundle branch pacing (high thresholds (>3.5V / 1ms); no left bundle branch pacing criteria; no left bundle branch correction).
  Electrocardiographic optimization allowed in order to obtain the narrowest QRS.
  Interventions: Procedure: Conduction system pacing
- Biventricular pacing (Active Comparator): Pacing from the right ventricular and coronary sinus lead. Electrocardiographic optimization with fusion-optimized intervals (FOI).
  Crossover from biventricular pacing to conduction system pacing will be allowed in the following situations: coronary sinus cannot be cannulated; no lateral or posterolateral branches; or phrenic stimulation.
  Interventions: Procedure: Biventricular pacing

INTERVENTIONS:
Procedure: Conduction system pacing — Conduction system pacing implant as a Resynchronization therapy.
  Arms: Conduction system pacing
Procedure: Biventricular pacing — Biventricular pacing implant
  Arms: Biventricular pacing

SUMMARY:
Conduction system pacing vs biventricular resynchronization therapy in systolic dysfunction and wide QRS: mortality, heart failure hospitalization or cardiac transplant (CONSYST-CRT II trial).

Superiority trial that aims to study the composite endpoint consisting of all-cause mortality, cardiac transplant or heart failure hospitalization at 12-month follow-up.

DETAILED DESCRIPTION:
To date, studies have shown that conduction system pacing could get similar clinical and echocardiographic responses to those obtained with biventricular therapy.

This study will randomize 320 patients to a strategy of biventricular pacing versus conduction system pacing.

CONSYST-CRT II study will analyze a clinical endpoint as primary endpoint and the following parameters in both groups: left ventricular ejection fraction, ventricular volumes, echocardiographic response (>=15% decrease in left ventricular end-systolic volume), NYHA functional class, heart failure hospitalization, all-cause mortality, cardiac transplant, QRS shortening, echocardiographic dyssynchrony (atrioventricular, interventricular, intraventricular) and global longitudinal strain.

As a secondary endpoint, baseline predictors of response to conduction system pacing and biventricular pacing according to cardiac magnetic ressonance and electrocardiographic imaging will be studied.

Clinical, electrocardiographic, echocardiographic follow-up will be performed during 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient must indicate acceptance to participate in the study by signing an informed consent document.
* Patient must be ≥ 18 years of age.
* Left bundle branch block, QRS ≥130 and LVEF <=35%. No indication of stimulation for AV block.
* Non-left bundle branch block, QRS ≥150 and LVEF <=35%.
* Resynchronization therapy indication for ventricular dysfunction (LVEF <40%) and indication of cardiac pacing for AV block.
* LVEF <=35% in NYHA class III or IV, atrial fibrillation and intrinsic QRS >=130 ms, provided a strategy to ensure biventricular capture is in place.

Exclusion Criteria:

* Myocardial infarction, unstable angina or cardiac revascularization during the previous 3 months.
* Pregnancy.
* Participating currently in a clinical investigation that includes an active treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Composite end-point: all-cause mortality, cardiac transplant or heart failure hospitalization. | 1 year
  Clinical follow-up at 12 months

SECONDARY OUTCOMES:
Change in left ventricular ejection fraction. | 6 months; 1 year
  Left ventricular ejection fraction measured with Simpson method with echocardiography.
Change in left ventricular end-systolic volume. | 6 months; 1 year
  Left ventricular volumes measured with echocardiography. Simpson rule from 2- and 4-chamber apical views.
Echocardiographic response. | 6 months; 1 year
  >=15% decrease in left ventricular end-systolic volume
Change in NYHA functional class. | 6 months; 1 year
  NYHA functional class I, II, III, or IV
QRS shortening. | Immediately after the intervention
  QRS duration (milliseconds). QRS onset measured from fast deflection and from spike.
Correction of septal flash. | 15 days; 6 months; 1 year
  Fast inward-outward movement of the interventricular septum in early systole. Using M-mode in parasternal short and long-axis views, septal flash was quantified (in millimeters) as the highest amplitude of the early inward motion measured from the resting position prior to the onset of septal contraction. The pair of septal flash measures (baseline and final) was obtained at the axis with the highest baseline SF.
Correction of auriculoventricular dyssynchrony. | 15 days; 6 months; 1 year
  Left ventricular filling time. The left ventricular filling time was measured from the onset of the E-wave to the end of the A-wave, and the R-R interval was measured to calculate the percentage of filling time relative to the cardiac cycle (LV filling time/RR, %).
Correction of interventricular dyssynchrony. | 15 days; 6 months; 1 year
  Quantified using pulsed Doppler and calculated as the time difference between QRS onset and the onset of the flow wave in the right and left outflow tracts.
Change in global longitudinal strain (GLS). | 15 days; 6 months; 1 year
  Strain myocardial deformation of the left ventricle was quantified offline from 2-dimensional echocardiography using speckle tracking (2Dstrain, Echo Pac, version 202.41.0, GE Healthcare Milwaukee, WI). The long-axis cine images (2-, 3-, and 4-chamber views), were used to determine GLS.
Description of baseline predictors of response to conduction system pacing and biventricular pacing. Cardiac fibrosis quantification. | Baseline (pre intervention).
  Cardiac fibrosis quantification (grams of fibrosis)
Description of baseline predictors of response to conduction system pacing and biventricular pacing with Electrocardiographic Imaging. Left ventricular activation time (LVAT), ms. | Baseline (pre intervention). And immediately after the intervention
  Left ventricular activation time (LVAT), ms.
Description of baseline predictors of response to conduction system pacing and biventricular pacing with Electrocardiographic Imaging. Ventricular electrical uncoupling (VEU). | Baseline (pre intervention). And immediately after the intervention
  Ventricular electrical uncoupling (VEU) = mean left ventricular activation time - mean right ventricular activation time, ms
Description of baseline predictors of response to conduction system pacing and biventricular pacing with Electrocardiographic Imaging. Left ventricular dyssynchrony index (LVDI). | Baseline (pre intervention). And immediately after the intervention
  Left ventricular dyssynchrony index (LVDI): standard deviation of individual activations recorded from the left ventricle.
Description of baseline predictors of response to conduction system pacing and biventricular pacing with Electrocardiographic Imaging. Conduction velocity (cm/s). | Baseline (pre intervention). And immediately after the intervention
  Conduction velocity (cm/s).

CONTACTS AND LOCATIONS:
Overall Officials: José Mª Tolosana, MD, PhD, Principal Investigator — Hospital Clínic de Barcelona. Institut d'Investigacions Biomèdiques August Pi i Sunyer; Margarida Pujol López, MD, Principal Investigator — Hospital Clínic de Barcelona. Institut d'Investigacions Biomèdiques August Pi i Sunyer; Lluís Mont, MD, PhD, Study Chair — Hospital Clínic de Barcelona. Institut d'Investigacions Biomèdiques August Pi i Sunyer
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No